CLINICAL TRIAL: NCT00289315
Title: LA Health: A Prospective Study of Primary and Secondary Obesity Prevention in Children and Adolescents
Brief Title: The Louisiana (LA) Health Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Corby K. Martin, Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LA Health; R01HD048483-01 (NIH)
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Environment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Primary (Environmental) Prevention of Weight Gain
  Interventions: Behavioral: Primary (Environmental) Weight Gain Prevention
- Arm 2 (Experimental): Primary (Envrironmental) and Secondary (Behavioral) Weight Gain Prevention Program
  Interventions: Behavioral: Primary (Environmental) Weight Gain Prevention; Behavioral: Secondary (Behavioral) Weight Gain Prevention
- Arm 3 (Experimental): Control - no Environmental or Behavioral Program intervention
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Primary (Environmental) Weight Gain Prevention — School-based program that modifies the school environment to promote healthy eating and physical activity
  Arms: Arm 1; Arm 2
Behavioral: Secondary (Behavioral) Weight Gain Prevention — School-based environmental program to promote healthy eating and physical activity in the overweight students.
  Arms: Arm 2
Behavioral: Control — Control program that does not include an active intervention for promoting healthy eating and physical activity.
  Arms: Arm 3

SUMMARY:
There is a worldwide pandemic of obesity with far-reaching consequences for the health of our nation. Obesity is the second leading cause of preventable death in the United States. Prevention of obesity, especially in children, has been deemed by public health policy makers to be one of the most important objectives for our country.

DETAILED DESCRIPTION:
There is a worldwide pandemic of obesity with far-reaching consequences for the health of our nation. Obesity is the second leading cause of preventable death in the United States. Prevention of obesity, especially in children, has been deemed by public health policy makers to be one of the most important objectives for our country. Obesity disproportionately affects citizens of minority and low socioeconomic status. A consensus of opinion has formed that the recently observed increased prevalence of obesity is caused by environmental and behavioral factors that favor easy access to high calorie foods and sedentary behavior. This prevention project, called LA Health, will test whether modification of these environmental and behavioral factors can prevent inappropriate weight gain in children who are enrolled in the fourth to sixth grades during Year 1. The primary aims of the LA Health project are to test the efficacy of two school-based approaches for obesity prevention. The two approaches are derived from two NIH-funded pilot studies called the HIPTeens project (a secondary prevention program) and the Wise Mind project (a primary prevention program). The study will test the efficacy of primary prevention alone and a combination of primary and secondary prevention in comparison to a no-treatment control group using a cluster randomization research design, with 18 school clusters from 9 different parishes randomly assigned to the three treatment arms. The following parishes were selected for the project: East Carroll, Madison, Franklin, East Feliciana, St. John, St. Helena, Pointe Coupee, Avoyelles, and Sabine Parishes. Thus far East Carroll, East Feliciana, St. John, Pointe Coupee, and Avoyelles Parishes have agreed to participate. We anticipate adding additional parishes in the second year of the project.The project will collaborate with a USDE funded project, LA GEAR UP, to test the relative efficacy obesity prevention programs for children who come from economically disadvantaged environments. The LA GEAR UP program is designed to enhance educational achievement. Since LA GEAR UP will be implemented in all 18 school clusters, all of the preventions intervention arms, including no-treatment, will be combined with an academic enhancement program. The study will span three years and will provide critical tests of strategies that modify the child's environment as a primary prevention strategy and provide health behavior modification via classroom instruction and internet counseling as a secondary prevention strategy. The study will also recruit a similar (but smaller) sample of students to measure changes in body weight relative to height, gender, and age over the same three-year period. This observation only control group will be studied to evaluate secular trends in changes in body weight so that body weight changes observed in the randomized trial can be interpreted within the context of stable versus unstable population changes in body weight. The results of this investigation will significantly impact public health policy related to obesity prevention in rural communities, minority communities, and in children from families that are economically disadvantaged.

ELIGIBILITY:
Inclusion Criteria:

* Being one of the LA GEAR UP middle schools or a feeder elementary school
* Having an enrollment of at least 100 students per school
* All students in grades 4-6 of participating schools

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2060 (Actual)
Dates: Start 2005-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Williamson DA, Han H, Johnson WD, Martin CK, Newton RL Jr. Modification of the school cafeteria environment can impact childhood nutrition. Results from the Wise Mind and LA Health studies. Appetite. 2013 Feb;61(1):77-84. doi: 10.1016/j.appet.2012.11.002. Epub 2012 Nov 12. PMID 23154216
- [Derived] Williamson DA, Champagne CM, Harsha DW, Han H, Martin CK, Newton RL Jr, Sothern MS, Stewart TM, Webber LS, Ryan DH. Effect of an environmental school-based obesity prevention program on changes in body fat and body weight: a randomized trial. Obesity (Silver Spring). 2012 Aug;20(8):1653-61. doi: 10.1038/oby.2012.60. Epub 2012 Mar 8. PMID 22402733
- [Derived] Newton RL, Thomson JL, Rau KK, Ragusa SA, Sample AD, Singleton NN, Anton SD, Webber LS, Williamson DA. Psychometric characteristics of process evaluation measures for a rural school-based childhood obesity prevention study: Louisiana Health. Am J Health Promot. 2011 Jul-Aug;25(6):417-21. doi: 10.4278/ajhp.090914-ARB-297. PMID 21721969
- [Derived] Newton RL, Han H, Sothern M, Martin CK, Webber LS, Williamson DA. Accelerometry measured ethnic differences in activity in rural adolescents. J Phys Act Health. 2011 Feb;8(2):287-95. doi: 10.1123/jpah.8.2.287. PMID 21415456
- [Derived] Williamson DA, Han H, Johnson WD, Stewart TM, Harsha DW. Longitudinal study of body weight changes in children: who is gaining and who is losing weight. Obesity (Silver Spring). 2011 Mar;19(3):667-70. doi: 10.1038/oby.2010.221. Epub 2010 Sep 30. PMID 20885393
- [Derived] Martin CK, Thomson JL, LeBlanc MM, Stewart TM, Newton RL Jr, Han H, Sample A, Champagne CM, Williamson DA. Children in school cafeterias select foods containing more saturated fat and energy than the Institute of Medicine recommendations. J Nutr. 2010 Sep;140(9):1653-60. doi: 10.3945/jn.109.119131. Epub 2010 Jul 28. PMID 20668251
- [Derived] Gabriele JM, Stewart TM, Sample A, Davis AB, Allen R, Martin CK, Newton RL Jr, Williamson DA. Development of an internet-based obesity prevention program for children. J Diabetes Sci Technol. 2010 May 1;4(3):723-32. doi: 10.1177/193229681000400328. PMID 20513340
- [Derived] Williamson DA, Champagne CM, Han H, Harsha D, Martin CK, Newton RL, Ryan DH, Sothern MS, Stewart TM, Webber LS. Increased obesity in children living in rural communities of Louisiana. Int J Pediatr Obes. 2009;4(3):160-5. doi: 10.1080/17477160802596148. PMID 19089707
- [Derived] Williamson DA, Champagne CM, Harsha D, Han H, Martin CK, Newton R Jr, Stewart TM, Ryan DH. Louisiana (LA) Health: design and methods for a childhood obesity prevention program in rural schools. Contemp Clin Trials. 2008 Sep;29(5):783-95. doi: 10.1016/j.cct.2008.03.004. Epub 2008 Mar 26. PMID 18448393

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1-Primary Prevention of Weight Gain: Primary Prevention of weight gain
  Primary weight gain prevention: School-based program that modifies the school environment to promote healthy eating and physical activity
  Primary Prevention: School-based environmental program to promote healthy eating and physical activity.
- Arm 2-Primary and Secondary Weight Gain Prevention Program: Primary and secondary weight gain prevention program
  Primary and Secondary Prevention: School-based program that combines an environmental weight gain prevention program with a curriculum/internet-based program to promote weight loss in overweight students
- Arm 3-Control: Control
  Control: Control program that does not include an active intervention for promoting healthy eating and physical activity.
Period: Overall Study
Arm/Group | Arm 1-Primary Prevention of Weight Gain | Arm 2-Primary and Secondary Weight Gain Prevention Program | Arm 3-Control
Started | 713 | 760 | 587
Completed | 612 | 638 | 447
Not Completed | 101 | 122 | 140

BASELINE CHARACTERISTICS:
Population: Only participants with complete data (baseline and at least one of two follow-up measurements) were included in the analysis.
Groups:
- Arm 1: Primary Prevention of weight gain
  Primary weight gain prevention: School-based program that modifies the school environment to promote healthy eating and physical activity
  Primary Prevention: School-based environmental program to promote healthy eating and physical activity.
- Arm 2: Primary and secondary weight gain prevention program
  Primary and Secondary Prevention: School-based program that combines an environmental weight gain prevention program with a curriculum/internet-based program to promote weight loss in overweight students
- Arm 3: Control
  Control: Control program that does not include an active intervention for promoting healthy eating and physical activity.
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 704 | 725 | 586 | 2015
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.5 (1.2) | 10.5 (1.2) | 10.6 (1.2) | 10.5 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 412 | 413 | 351 | 1176
  Male | 292 | 312 | 235 | 839

OUTCOME MEASURES:

1. Primary Outcome: % Body Fat (Boys)
Description: change in percent body fat between Baseline and 3 years for boys
Time Frame: Baseline and 3 years
Population: children in primary prevention, primary + secondary prevention, and control group (boys)
Measure: Mean (Standard Error); unit: percentage of body fat
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 292 | 312 | 235
percentage of body fat | -1.3 (0.59) | -2.0 (0.54) | -0.11 (0.68)

2. Primary Outcome: BMI Z-score (Boys)
Description: Body mass index z-scores are measures of relative weight adjusted for child age and sex. The Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to the mean. Negative numbers indicate BMI values lower than the mean and positive numbers indicate BMI values higher than the mean
Time Frame: Baseline and three years
Population: primary preventions, primary + secondary prevention, control group (boys)
Measure: Mean (Standard Error); unit: z score
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 292 | 312 | 235
z score | 0.022 (0.033) | 0.01 (0.03) | 0.055 (0.04)

3. Primary Outcome: % Body Fat (Girls)
Description: change in percent body fat between Baseline and 3 years for girls
Time Frame: Baseline and 3 years
Population: children in primary prevention, primary + secondary prevention, and control group (girls)
Measure: Mean (Standard Error); unit: percentage of body fat
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 412 | 413 | 351
percentage of body fat | 2.8 (.34) | 3.0 (0.32) | 3.9 (0.39)

4. Primary Outcome: BMI Z-score (Girls)
Description: as for outcome 2
Time Frame: Baseline and three years
Population: primary preventions, primary + secondary prevention, control group (girls)
Measure: Mean (Standard Error); unit: z score
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 412 | 413 | 351
z score | .017 (.021) | .069 (.021) | .076 (.025)

ADVERSE EVENTS:
Time Frame: Three years
Arm/Group | Arm 1 | Arm 2 | Arm 3
All-Cause Mortality (participants affected / at risk) | 0/713 | 0/760 | 0/587
Serious Adverse Events (participants affected / at risk) | 0/713 | 0/760 | 0/587
Other Adverse Events (participants affected / at risk) | 0/713 | 0/760 | 0/587

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No